CLINICAL TRIAL: NCT04435990
Title: Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled, Efficacy and Safety Clinical Trial With SCIT in Patients With Rhinitis/Rhinoconjunctivitis With or Without Mild to Moderate Asthma Sensitized to Dpt. and/or D. Farinae
Brief Title: Efficacy and Safety Evaluation for the Treatment of Allergy Against Mites
Acronym: MM09-SIT-023
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Collaborators: BioClever 2005 S.L. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MM09-SIT-023; 2018-004262-34 (EudraCT Number)
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Rhinitis, Allergic; Rhinoconjunctivitis; Asthma, Allergic
Keywords: Rhinitis/ Rhinoconjunctivitis; Mild to moderate asthma; Allergy; Immunotherapy; Mites
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multi centre, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the trial, both the investigator and the included subjects will be unaware of the treatment each subject is receiving.
  The person in charge of data analysis will also not know the treatment assigned to each subject until the database has been closed.
  So that neither the subject nor the investigator knows what treatment each subject is receiving, all the trial medication is identical in terms of outer packaging and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental:10,000 MM09 (Experimental): 10,000 TU/mL of subcutaneous immunotherapy
  Interventions: Biological: 10,000 MM09
- Experimental: 30,000 MM09 (Experimental): 30,000 TU/mL of subcutaneous immunotherapy
  Interventions: Biological: 30,000 MM09
- Placebo subcutaneous (Placebo Comparator): The same solution and presentation as the active treatment, but without any active ingredients.
  Interventions: Biological: Placebo subcutaneous

INTERVENTIONS:
Biological: 10,000 MM09 — Purified allergenic extract, and adsorbed in aluminum hydroxide and polymerized with glutaraldehyde, mite mixture (Dermatophagoides pteronyssinus and Dermatophagoides farinae) with a concentration of 10,000 UT / mL
  Arms: Experimental:10,000 MM09
Biological: 30,000 MM09 — Purified allergenic extract, and adsorbed in aluminum hydroxide and polymerized with glutaraldehyde, mite mixture (Dermatophagoides pteronyssinus and Dermatophagoides farinae). The concentration is 30,000 UT / mL
  Arms: Experimental: 30,000 MM09
Biological: Placebo subcutaneous — The same solution and presentation as the active treatment, but without active ingredients.
  Arms: Placebo subcutaneous

SUMMARY:
A double-blinded, placebo-controlled, prospective, multicenter randomized of 2 active treatment groups, compared to 1 placebo group, for the determination of the efficacy and safety of subcutaneous immunotherapy in patients with rhinitis/rhinoconjunctivitis with or without asthma, sensitised to Dermatophagoides pteronyssinus and /or Dermatophagoides farinae.

DETAILED DESCRIPTION:
Double blind, multicenter, parallel placebo controlled study. It includes 150 subjects sensitised to mites, from 12 to 65 years of age. Medication treatment of 1 year. The main outcome: CSMS

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age between 12 and 65, both genders.
* Subjects with a confirmed clinical history of inhalant allergy (intermittent or persistent moderate-severe rhinitis and/or rhinoconjunctivitis according to the ARIA classification with or without intermittent or persistent mild-moderate controlled asthma according to the GEMA 5.0 definition) caused by allergy to Dermatophagoides pteronyssinus and/or Dermatophagoides farinae. The diagnosis of asthma will be valid from 12 months prior to signing the informed consent.
* Subjects with a positive skin prick-test wheal size >5 mm higher diameter due to Dermatophagoides pteronyssinus and/or Dermatophagoides farinae. The positive and negative control of the test should give consistent results. The results will be valid 12 months prior to the signing of the informed consent.
* Specific immunoglobulin E against house dust mites >3,5 KU/mL (InmunoCAP® o Immulite), for the complete extract of Dermatophagoides pteronyssinus and / or for Dermatophagoides farinae or for some of the molecular components of these allergenic sources
* Subjects should preferably be monosensitized to the study allergens. In case of subjects sensitized to other aeroallergens, only those with the following characteristics may be included in the study:

  * Subjects with positive skin test to Blomia tropicalis and Lepidoglyphus destructor, whose specific IgE values do not exceed or equal the values for the study allergens. The maximum specific IgE value for these allergens is 3.5 KU/L.
  * Subjects with positive skin tests to epithelia, as long as they present occasional exposure and symptomatology.
  * Subjects with positive skin tests to pollens, whose specific IgE values do not exceed or equal the values of the allergens in the study and who do not present exacerbations during the pollen season. The maximum value of specific IgE for these allergens is 17.5 KU/L.
* Subjects with negative skin test for fungi
* Women of childbearing age (from menarche) must present a urine pregnancy test with a negative result at the time of joining the trial, before the first administration of the IMP.
* Women of childbearing age participating in the trial must agree to use an appropriate method of contraception, meaning any act, device, or medication to prevent conception or viable pregnancy, during the trial if they are sexually active.
* Subjects with a diagnosis of asthma according to the GEMA 5.0 guideline.
* Subjects capable of complying with the dosing regimen.
* Subjects who own an smartphone for symptom registration and medication

Exclusion Criteria:

* Subjects who have received previous immunotherapy in the previous 5 years to dander, fungi, and mites.
* Subjects in whom immunotherapy may be subject to an absolute general contraindication according to the criteria of the Immunotherapy Committee of the Spanish Society of Allergy and Clinical Immunology and the European Allergy and Clinical Immunology Immunotherapy Subcommittee.
* Subjects with persistent severe or uncontrolled asthma, with an FEV1<70% of baseline despite adequate pharmacological treatment at the time of inclusion in the trial. Also subjects with intermittent or persistent rhinitis/rhinoconjunctivitis with severe symptoms in whom oral or systemic antihistamine therapy is contraindicated.
* Subjects who have previously presented a serious secondary reaction during the performance of diagnostic skin tests using the prick test.
* Subjects under treatment with β-blockers.
* Clinically unstable subjects at the time of inclusion in the trial (acute asthma exacerbation, respiratory infection, feverish process, acute urticaria, etc.).
* Subjects with chronic active urticaria, severe dermographism, severe atopic dermatitis, sunburn, active psoriasis with lesions in areas where skin prick test will be performed, or a history of hereditary angioedema.
* Subjects with any other disease not related to moderate rhinoconjunctivitis or asthma, but of potential severity and that may interfere with treatment and follow-up (epilepsy, psychomotor impairment, uncontrolled diabetes, malformations, multiple surgeries, nephropathy).
* Subjects with autoimmune disease (thyroiditis, lupus, etc.), tumor diseases or with a diagnosis of immunodeficiencies.
* Subject whose condition prevents him/her from offering cooperation and/or who has serious mental illness.
* Subjects with a known allergy to other components of the investigational medicinal product other than the allergen.
* Subjects with diseases of the lower respiratory tract other than asthma such as emphysema or bronchiectasis.
* Direct investigator's relatives.
* Pregnant women or breastfeeding women.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CSMS: Combined Symptoms and Medication Score | 12 months
  Evaluation of the number of symptoms and the consumption of medication for symptoms rhinitis / rhinoconjunctivitis of each subject during the trial, of the groups with each other and with respect to placebo.

SECONDARY OUTCOMES:
Medication-free days | 12 months
  Number of days that the subjects need no medication
Symptom-free days | 12 months
  Number of days that the subjects have no symptom
Number of participants with treatment-related adverse events as assessed by MM09-SIT-023 | 12 months
  Comparison between the beginning and end of the trial and among active groups and placebo
Quality of life associated with asthma | 12 months
  The quality of life associated with asthma will be measured following the GINA questionnaire.
  The GINA questionnaire consists of 4 questions. In questions 1-4, patients recall their experience during the last 4 weeks and answer using YES or NO.
  The interpretation of the answers is as follows:
  Well-controlled: None of the answers are YES Partly controlled: 1 - 2 answers are YES Uncontrolled: 3-4 answers are YES
Quality of life associated with rhinitis | 12 months
  The quality of life associated with rhinitis will be measured following the test ESPRINT-15.
  The scoring of the questionnaire will be carried out as follows: The global sum of the scores (ranging from "0 = nothing has bothered me" to "6 = it has bothered me a lot") of the 14 items plus the score given in the general questionnaire (ranging from "0 = Excellent" to "4 = Bad"). This sum is divided by the total number of items (15 items).
  The interpretation of the scores is between 0 (low impact) and 6 (high impact).
Visual Analogue Scale (VAS) | 12 months
  Visual Analogue Scale in which the subject has to indicate how he/she feels regarding to his allergy symptoms at the moment from 1 to 10. Being 1 very bad and 10 very well.
Immunological parameters | 12 months
  Analyses of total IgE and specific IgA,IgG and IgG4

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Moreno, MD, Study Director — Centro Médico ASISA
Locations (32):
- Spain (32):
  - Hospital Provincial de Conxo, Santiago de Compostela, A Coruña
  - IMED Elche, Elche, Alicante
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante
  - Clinica Tecma, Valencia, Alzira
  - Clinica Virgen del Rosario, Algeciras, Cadiz
  - Hospital HLA Jerez Puerta Sur, Jerez de la Frontera, Cádiz
  - Hospital Dr. Peset, Valencia, España
  - Hospital General Universitario Santa Maria de Rosell, Cartagena, Murcia
  - Hospital Rivera Povisa, Vigo, Pontevedra
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario San Juan de Alicante, Alicante
  - Clínica Dermatológica y Alergia, Badajoz
  - Hospital Quironsalud Clideba, Badajoz
  - Hospital Sant Pere Claver, Barcelona
  - Clínica Corachan, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Cenvi Medic, Barcelona
  - Allergocenter, Barcelona
  - Clinica privada, Bilbao
  - Centro Médico ASISA Dr. Lobatón, Cadiz
  - Centro Médico Puerto, Cadiz
  - Hospital Quiron Salud Córdoba, Córdoba
  - Hospital Polusa, Lugo
  - Clinica privada, Málaga
  - Hospital Comarcal de Melilla, Melilla
  - Clinica Privada, Murcia
  - Alergocantabria, Santander
  - Hospital Quiron Infanta Luisa, Seville
  - Clinica Lanuza, Valencia
  - Hospital Universitario Y Politecnico La Fe, Valencia
  - Clinica IMED, Valencia
  - Hospital de Sagunto, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piacentini GL, Vicentini L, Mazzi P, Chilosi M, Martinati L, Boner AL. Mite-antigen avoidance can reduce bronchial epithelial shedding in allergic asthmatic children. Clin Exp Allergy. 1998 May;28(5):561-7. doi: 10.1046/j.1365-2222.1998.00260.x. PMID 9645592
- [Background] Yepes-Nunez JJ, Gomez C, Espinoza Y, Cardona R. [The impact of subcutaneous immunotherapy with Dermatophagoides farinae and Dermatophagoides pteronyssinus on the quality of life of patients with allergic rhinitis and asthma]. Biomedica. 2014 Apr-Jun;34(2):282-90. doi: 10.1590/S0120-41572014000200014. Spanish. PMID 24967933
- [Background] Cardona R, Lopez E, Beltran J, Sanchez J. Safety of immunotherapy in patients with rhinitis, asthma or atopic dermatitis using an ultra-rush buildup. A retrospective study. Allergol Immunopathol (Madr). 2014 Mar-Apr;42(2):90-5. doi: 10.1016/j.aller.2012.07.005. Epub 2012 Dec 20. PMID 23265265
- [Background] Bousquet J, Hejjaoui A, Clauzel AM, Guerin B, Dhivert H, Skassa-Brociek W, Michel FB. Specific immunotherapy with a standardized Dermatophagoides pteronyssinus extract. II. Prediction of efficacy of immunotherapy. J Allergy Clin Immunol. 1988 Dec;82(6):971-7. doi: 10.1016/0091-6749(88)90133-9. PMID 3204255
- [Background] Branco Ferreira M, Spinola Santos A, Pereira Santos MC, Palma Carlos ML, Pereira Barbosa MA, Palma Carlos AG. Efficacy and safety of specific immunotherapy with a modified mite extract. Allergol Immunopathol (Madr). 2005 Mar-Apr;33(2):80-5. doi: 10.1157/13072918. PMID 15808114